CLINICAL TRIAL: NCT04515862
Title: A Randomızed Controlled Study On Analysıs Of Effect Of Hospıtal Based Breast-Feedıng Group Traınıng Provıded In Early Postpartum Perıod About Breast-Feedıng Self-Effıcacy And Breast-Feedıng Status Of Maternals
Brief Title: Hospital-Based Breastfeeding Training İn The Early Postpartum Period
Acronym: BF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, YEŞİM YEŞİL, Research Assistant, Ege University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Yesim Yesil
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Postpartum; Women; Education
Keywords: Breastfeeding; group training; Self-Effıcacy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: The study was applied to mothers who gave birth at a time when they felt well after being taken to their postnatal room. First, the mothers who met the inclusion criteria were informed, after obtaining written consent, the mothers were randomized using a random number table and then assigned to the intervention and control groups.
  All mothers were asked to fill in the breastfeeding self-efficacy scale form together with the questionnaire before the intervention. Later, a training program was conducted in the hospital with the mothers in the intervention group.
  In the data collection phase of the study, 1180 women were evaluated in terms of sampling criteria. 1152 women (who did not meet the criteria or refused to participate) were excluded from the study. 90 randomized women were divided into two groups as intervention and control group. During the follow-up, 5 women in the intervention group and 5 women in the control group were excluded from the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Intervention group: Mothers in the intervention group were included in the breastfeeding training program with the group training method. The training program was developed by the researchers, and the content of the program was evaluated with the expert opinion of academicians, obstetricians, nurses and breastfeeding counselor midwives working on breastfeeding.
  Interventions: Other: Breastfeeding education
- control (No Intervention): Control Group:Routine obstetric care and treatment procedures were applied to the mothers in the control group. In the hospital where the study was conducted, all mothers are routinely evaluated for breastfeeding by an infant nurse.

INTERVENTIONS:
Other: Breastfeeding education — The importance of breastfeeding Benefits of breastfeeding for mother and baby Structure of the breast and milk production Breastfeeding techniques and positions Breastfeeding problems and breast care
  Arms: intervention

SUMMARY:
H1: "Breastfeeding Self-Efficacy Status" is higher in mothers who received postnatal hospital-based breastfeeding group training compared to the control group receiving routine care.

H2: The level of knowledge obtained according to the "Pre-test Post-test Question Form" in mothers who received postnatal hospital-based breastfeeding group training is higher than before the education.

H3: The status of starting and successfully continuing breastfeeding is higher in mothers who received postnatal hospital-based breastfeeding group training compared to the control group who received routine care.

DETAILED DESCRIPTION:
Follow-up data of all mothers were collected by phone at 4 and 12 weeks. For this reason, the phone numbers of the mothers and a relative were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Can be contacted,
2. had a single birth,
3. Those who are 18 years old or older,
4. Residing in Izmir,
5. able to use phone
6. were determined to be mothers with no health problems in the mother and the baby

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — breastfeeding education was given to women
Enrollment: 80 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-01-30 (Actual); Study Completion 2016-03-15 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale | twelve weeks
  This scale was developed by Cindy-Lee Dennis to measure breastfeeding competence and consists of 2 subscales and 33 items. The Turkish validity and reliability of the breastfeeding proficiency scale was made by Ekşioğlu and Çeber (2011). Breastfeeding self-efficacy increases as the total score increases in the 5-point Likert-type scale with a Cronbach Alpha coefficient of 0.91. The lowest score is 33, the highest score is 165.
Pre-Test Post-Test Information Form | twelve weeks
  It is a question form consisting of 25 questions in order to evaluate the knowledge about breastfeeding and breast milk before and after the training. The first application was done before the training and the second application was carried out in the 12th week.
Breastfeeding levels of mothers | four weeks, twelve weeks
  The exclusive breastfeeding levels of their babies in the fourth and twelfth weeks of the mothers who received and did not receive education were evaluated.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Binns C, Lee M, Low WY. The Long-Term Public Health Benefits of Breastfeeding. Asia Pac J Public Health. 2016 Jan;28(1):7-14. doi: 10.1177/1010539515624964. PMID 26792873
- [Background] Yilmaz M, Aykut M. The effect of breastfeeding training on exclusive breastfeeding: a randomized controlled trial. J Matern Fetal Neonatal Med. 2021 Mar;34(6):925-932. doi: 10.1080/14767058.2019.1622672. Epub 2019 Jul 25. PMID 31345049
- [Background] Eksioglu AB, Ceber E. Translation and validation of the Breast-feeding Self-efficacy Scale into Turkish. Midwifery. 2011 Dec;27(6):e246-53. doi: 10.1016/j.midw.2010.10.009. Epub 2010 Dec 8. PMID 21145148